CLINICAL TRIAL: NCT05963568
Title: Stroke Minimization Through Additive Anti-atherosclerotic Agents in Routine Treatment II Study (SMAART II)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Northern California Institute of Research and Education (Other)
Responsible Party: Principal Investigator, Bruce Ovbiagele, Chief of Staff, Northern California Institute of Research and Education
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22-37310
Record Dates: First submitted 2022-08-11; First posted 2023-07-27 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Medication Adherence
MeSH Terms: conditions — Stroke; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients allocated to the experimental arm will receive Two (2) (Polycap ®) taken orally once a day. A capsule of Polycap ® contains 100mg of Aspirin, 20mg of simvastatin, 12.5mg hydrochlorothiazide, 5mg of ramipril and 50mg of atenolol. Patients assigned to Polypill will have their antihypertensive agents, lipid modifiers and anti-thrombotic agents withdrawn & replaced with the Polypill if they are already receiving such treatments before enrollment.
  Interventions: Drug: Polycap
- Control arm (No Intervention): Patients allocated to the usual care arm will receive standard of care therapies for secondary prevention with drugs and doses left at the discretion of the treating physicians. Since our focus is to isolate the effect of the polypill strategy itself & create equipoise, at study inception providers for patients in both study arms will receive a brief one-time (Skype-based) training & a one time email synopsis on guideline recommended biomarker targets after stroke.

INTERVENTIONS:
Drug: Polycap — Patients allocated to the experimental arm will receive Two (2) (Polycap ®) taken orally once a day. A capsule of Polycap ® contains 100mg of Aspirin, 20mg of simvastatin, 12.5mg hydrochlorothiazide, 5mg of ramipril and 50mg of atenolol. Patients assigned to Polypill will have their antihypertensive agents, lipid modifiers and anti-thrombotic agents withdrawn and replaced with the Polypill if they are already receiving such treatments before enrollment.
  Arms: Intervention

SUMMARY:
The overall objective of the Stroke Minimization through Additive Anti-atherosclerotic Agents in Routine Treatment II (SMAART-II) is to deploy a hybrid study design to firstly, demonstrate the efficacy of a polypill (Polycap ®) containing fixed doses of antihypertensives, a statin, and antiplatelet therapy taken as two capsules, once daily orally in reducing composite vascular risk over 24 months vs. usual care among 500 recent stroke patients encountered at 12 hospitals in Ghana. Secondly, SMAART II seeks to develop an implementation strategy for routine integration and policy adoption of this polypill for post-stroke cardiovascular risk reduction in an under-resourced system burdened by suboptimal care and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Above the age of 18 years; male or female
* Ischemic stroke diagnosis no greater than two months before enrollment. Ischemic strokes including� lacunar, large-vessel atherosclerotic, cardio-embolic subtypes are eligible
* Subjects with stroke may present with at least one of the following additional conditions:

Documented diabetes mellitus or previous treatment with oral hypoglycemic or insulin; documented hypertension >140/90mmHg or previous treatment with antihypertensive medications; Mild to moderate renal dysfunction (eGFR 60-30ml/min/1.73m2); Prior myocardial infarction

* Legally competent to sign informed consent.

Exclusion Criteria:

* Unable to sign informed consent
* Contraindications to any of the components of the polypill
* Hemorrhagic stroke
* Severe cognitive impairment/dementia or severe global disability limiting the capacity of self-care
* Severe congestive cardiac failure (NYHA III-IV)
* Severe renal disease, eGFR <30ml/min/1.73m2), renal dialysis; awaiting renal transplant or transplant recipient
* Cancer diagnosis or treatment in past 2 years
* Need for oral anticoagulation at the time of randomization or planned in the future months;
* Significant arrhythmias (including unresolved ventricular arrhythmias or atrial fibrillation)
* Nursing/pregnant mothers
* Do not agree to the filing, forwarding and use of his/her pseudonymized data.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Composite vascular risk factor control | 12 and 24 months
  Proportion of people who have 0, 1, 2 and 3 of the following: systolic BP <140 mm Hg, LDL-cholesterol <100mg/dl, antiplatelet adherence by pill count >90%) at month 12 and month 24 (sustainment of effect)

SECONDARY OUTCOMES:
Major adverse cardiovascular events (MACE) | 24 months
  MACE to be assessed include recurrent stroke: fatal/severely disabling stroke or non-fatal stroke; coronary artery disease: acute STEMI/NSTEMI, sudden cardiac deaths. MACE will be confirmed by a blinded adjudication committee by reviewing available clinical notes supported by investigations for example CT scans, EKGs, troponin tests, death certificates or verbal autopsy if death occurs outside hospital.
Change in adherence to medical therapy | Month 3, 6, 9, 12, 18 & 24
Safety and tolerability | Up to 24 months
  Side effects, adverse events, treatment withdrawal
Health-related quality of life EuroQol-5D | Up to 24 months
  EuroQol-5D questionnaire (0-100 with 100 being the best)
Health-related quality of life Neuro-QoLTM | Up to 24 months
  NINDS Neuro-QoLTM (Quality of Life in Neurological Disorders) questionnaires (8-40 with 40 being the best)

OTHER OUTCOMES:
Organizational Capacity for Change Score | Up to 30 months
  Adoption i.e. Organizational Capacity for Change (OCC Scale Score comparison) with stratification by level of healthcare delivery. The measure is a 32-item multidimensional scale that evaluates an organization's capacity to upgrade or revise existing organizational competencies, while cultivating new competencies that enable the organization to survive and prosper. It comprises different aspects of leadership, employee behavior, and an organizational infrastructure supporting organizational change. Items are rated on a 5-point Likert scale. OCC has a Cronbach α of 0.87.
Mean Cost of Implementation | Up to 30 months
  Implementation Cost (mean monthly health expenses compared to standard of care)
Proportion who achieves systolic blood pressure <140 mmHg | Months 12 and 24
Proportion who achieves blood pressure <140/90 mmHg | Months 12 and 24
Proportion who achieves blood pressure < 130 / 80 mmHg | Months 12 and 24
Proportion who achieves LDL-cholesterol <100 mg/dl | Months 12 and 24
Proportion who achieves LDL-cholesterol <70 mg/dl | Months 12 and 24
Proportion who achieves antiplatelet adherence of at least >=80% | Months 12 and 24
Proportion who achieves antiplatelet adherence of at least >= 90% | Months 12 and 24
Comparison of absolute and mean changes from baseline for blood pressure | Up to 24 months
  systolic blood pressure, diastolic blood pressure, mean arterial blood pressure, measures of visit-to-visit variability in blood pressure
Comparison of absolute and mean changes from baseline for lipids | Up to 24 months
  Total cholesterol, LDL-cholesterol, HDL-cholesterol, and triglyceride
Proportion with recurrent strokes (fatal or non-fatal) | Up to 24 months
Proportion with coronary artery disease | Up to 24 months
Proportion with heart failure | Up to 24 months
Proportion with cardiovascular deaths | Up to 24 months
Proportion with all-cause mortality | Up to 24 months
Proportion with vascular cognitive impairment | Months 12 and 24
Proportion with treatment-limiting adverse drug reactions or side effects | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Kwame Nkrumah Institute of Science & Technology, Kumasi, Ghana